CLINICAL TRIAL: NCT07040904
Title: Mindfulness to Enhance Cognitive Health in Latinx Older Adults
Acronym: MLX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Todd Braver, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Tbraver
Record Dates: First submitted 2024-11-04; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Mindfulness; Alzheimer's Disease Related Dementia
Keywords: AD Biomarkers; Alzheimer's Disease; Alzheimer's disease and related dementias; cognitive behavioral intervention; Mindfulness; Mindfulness Training
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Randomization Description: After the pre-training assessment phase, participants will be randomized to either the Mindfulness Based Program or wait-list groups. The only difference between the two groups is that the wait-list group will not receive the mindfulness intervention until after they complete both pre- and post-assessments during the 4-month study period. Intervention Description: Mindfulness Program A novel and culturally-adapted version of the well-validated mindfulness-based stress reduction (MBSR) course will be used for the intervention. The adapted program curriculum embeds core MBSR principles and practices within a culturally responsive didactic framework developed directly from community focus-group feedback. The course will be delivered via a group meeting across 8 weeks, with weekly classes held at a local community center. All classes will be held in hybrid format, with most participants attending in person, but with a live-stream option offered via Zoom.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: mindfulness — MBSR: Mindfulness Program A novel and culturally-adapted version of the well-validated mindfulness-based stress reduction (MBSR) course will be used for the intervention. The adapted program curriculum embeds core MBSR principles and practices within a culturally responsive didactic framework developed directly from community focus-group feedback. The course will be delivered via a group meeting across 8 weeks, with weekly classes held at a local community center. All classes will be held in hybrid format, with most participants attending in person, but with a live-stream option offered via Zoom.

SUMMARY:
The primary objective of the proposed research is to investigate the promise and underlying mechanisms of mindfulness training as a preventative lifestyle intervention to enhance cognitive health in Latinx older adults, thereby mitigating risk of Alzheimer's Disease (AD) in a population that may be particularly vulnerable.

DETAILED DESCRIPTION:
This proposal rigorously examines the feasibility and mechanisms of action of a novel, culturally-sensitive mindfulness training program developed by the PIs, utilizing EEG methods and theoretically-optimized cognitive control tasks to assess neurocognitive effects. Additionally, blood-based assessment of AD biomarkers will be utilized to test whether biomarker status will moderate the effect of training, such that the neurocognitive benefits will be larger Latinx older adults with greater evidence of AD-related pathology. Furthermore, the study will also seek to elucidate the subjective effects of mindfulness training on daily-life experiences using ecological momentary assessment (EMA) methods. The study will utilize a mixed between and within-subject design involving longitudinal (pre vs. post-training) assessment and a wait-list control group. 60 Latinx older adults will first complete a baseline assessment protocol, followed by randomized assignment to either the mindfulness or wait-list group (N=30 in each group). The mindfulness group will receive 8 weeks of mindfulness training. During this 8-week period participants from both groups will also complete an EMA protocol, consisting of prompts occurring 4x/day on 3 random days per week, assessing subjective mindfulness states, practice experiences, mood, cognition, setting, and activity. Both groups will then return to repeat performance of the same assessment protocol. The assessment protocol involves two testing sessions performed on separate days, each involving completion of the Stroop and AX-CPT task while continuous EEG is recorded. The mindfulness training curriculum utilizes a novel adaptation of the well-validated mindfulness-based stress reduction (MBSR) course, that has been previously validated in focus groups. Participants will meet weekly with an instructor (either in-person or on-line) in classes to receive instructions and practice mindfulness skills. The curriculum embeds core MBSR principles and practices within a culturally-sensitive didactic framework, that includes four key modifications: (1) delivering all instruction in participants native Spanish language; (2) emphasizing/encouraging the connection between mindfulness practices and participants' personal religious beliefs (e.g., "connecting the breath/body to God"), (3) incorporating culturally unique experiences into group activities/exercises (e.g., sharing immigration stories and examining how alterations in perspective can influence meaning and affect), and (4) adding more familial focus to course content (e.g., highlighting how certain skills or practices can benefit the family). In addition to weekly class meetings, participants will also have access to instructional videos and guided audio practices available on their mobile device; on these devices, they will also be periodically prompted to partake in a short mindfulness behavioral task, a 2-minute breath-counting exercise. Finally, all participants will complete a blood draw at the end of the study to determine AD biomarker status. Outcomes will be assessed using EMA measures of daily mindfulness and mood/cognition as well as other qualitative self-report measures assessing the accessibility, utility and feasibility of the mindfulness training curriculum (Aim 1); EEG/ERP measures of state mindfulness and neurocognitive functioning (Aim 2); behavioral metrics of cognitive performance (Aim 2); and moderating role of AD biomarker status (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Hispanic/Latinx
* Age 65 and older
* Male, female, or non-binary
* Community living
* Medically stable and willing to undergo the study procedures
* No extensive mindfulness training experience

Exclusion Criteria:

* Clinically unstable psychiatric disorder that requires immediate treatment (e.g., ECT)
* Medical conditions suggesting significantly shortened lifespan (e.g., metastatic cancer) or prohibiting safe participation in the interventions/assessments (e.g., Parkinson's disease, musculoskeletal conditions)
* Sensory impairment (hearing, vision) preventing participation
* Current alcohol or substance abuse
* Current/concurrent cognitive training known to affect neuroplasticity (e.g., brain-training programs), or other interventions expected to affect neuroplasticity significantly (e.g., psychedelics, cholinesterase inhibitors, high-dose sedatives).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
EEG brain markers of cognitive functioning | Time-frame: 2 time-points - baseline/pre-intervention, and immediately after the intervention
  EEG indices of cognitive performances evoked by task stimuli and participant responses. ERP components of attention and cognitive control during task performance, focused on target-related P3 amplitude.
EEG brain markers of cognitive functioning | Time-frame: 2 time-points - baseline/pre-intervention, and immediately after the intervention
  EEG indices of cognitive performances evoked by task stimuli and participant responses. ERP components of attention and cognitive control during task performance, focused on cue-related Contingent Negative Variation (CNV).
AXCPT behavioral performance (reaction time) | Assessed at 2 timepoints: baseline/pre-intervention immediately post-intervention
  Behavioral performance indices during AXCPT task: AX-CPT - reaction time in milliseconds
AXCPT behavioral performance score (accuracy) | Assessed at 2 timepoints: baseline/pre-intervention immediately post-intervention
  Behavioral performance indices during AXCPT task: AX-CPT - % accuracy AX-CPT --% accuracy
Five Facet Mindfulness Questionnaire (FFMQ) score | Performed during the intervention (3x /week for 8 weeks)
  Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item self-report inventory used to measure five distinct facets of mindfulness. The five facets are observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience, each rated on a 5-point Likert scale.
The Mindful Attention Awareness Scale (MAAS) score | Performed during the intervention (3x /week for 8 weeks)
  The Mindful Attention Awareness Scale (MAAS) is a 15-item measure of mindfulness that prioritizes assessment of the general tendency to be attentive and aware of experiences in the present moment. It is is rated on a 6-point Likert scale (almost always, very frequently, somewhat frequently, somewhat infrequently, very infrequently, almost never).
Cognitive and Affective Mindfulness Scale (CAMS-R) score | Performed during the intervention (3x /week for 8 weeks)
  Cognitive and Affective Mindfulness Scale (CAMS-R) is used to evaluate symptoms of mindfulness as EMA (ecological momentary assessment) questions. It will be measured in a Likert scale (Not at all, Somewhat, Quite a bit, Almost completely)
Patient-Reported Outcomes Measurement Information System (Promis) score | Performed during the intervention (3x /week for 8 weeks)
  PROMIS (Patient-Reported Outcomes Measurement Information System) are item banks that measure common health outcomes across the domains of physical, mental, and social health.
National Institutes of Health Toolbox Emotion Battery (NIH-TOOLBOX-EB) score | baseline (pre-intervention) & immediately post-intervention
  National Institutes of Health Toolbox Emotion Battery for English- and Spanish-speaking adults (NIH-TOOLBOX-EB): National Institutes of Health Toolbox Emotion Battery for English- and Spanish-speaking adults (NIH-TOOLBOX-EB) A series of scales that will be rated on a 5-point Likert scale which include:
  1. General Life Satisfaction
  2. Meaning and Purpose
  3. Loneliness
  4. Sadness
  5. Positive Affect
  6. Fear Affect
  7. Perceived Stress
  8. Resilience Scale
  9. Sleep Quality Scale

SECONDARY OUTCOMES:
EEG metrics of mindfulness practice quality | Assessed at 2 timepoints: baseline/pre-intervention immediately post-intervention
  EEG spectral power (alpha, theta bands) evoked during guided mindfulness state induction

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the data collected in will be preserved through deposition in a public access data repository (i.e., Open Science Framework [OSF]). Raw self-report, transcription, and EMA data will be recoded, scored, and wrangled to "long" format to enhance accessibility and ease of use prior to sharing. All shared data will be deidentified.
Supporting Information: SAP, Analytic Code
Time Frame: Data will be made available one year after data collection begins and updated annually until the award period ends. All data, data wrangling procedures, registrations, and analysis scripts associated with published manuscripts will be organized into an easily accessible subfolder and made available no later than the time of publication acceptance. The data will be available for public access indefinitely, or until new guidelines are released regarding data archival duration.
Access Criteria: All data that is uploaded to OSF will be publicly available with no controlled access.